CLINICAL TRIAL: NCT05586295
Title: The Functional Evaluation on Antifatigue and Improving Sports Performance by Vitamin B Complex of BULIKELAO Sugar-coated Tablet
Brief Title: Vitamin B Complex Improved Exercise Performance and Anti-fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Collaborators: Prince Pharmaceutical Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Chi-Chang Huang, Distinguished Professor, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-037-A2
Record Dates: First submitted 2022-09-12; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Exercise Performance; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- EX plus (Experimental)
  Interventions: Other: EX plus

INTERVENTIONS:
Other: Placebo — Microcrystalline α-cellulose, shellac, calcium hydrogen phosphate, edible yellow No. 4, edible yellow No. 5, sucrose, silica, talc, oxidized starch, gelatin, magnesium stearate, palm wax.
  Arms: Placebo
Other: EX plus — Furanthiamine hydrochloride (vitamin B1), pyridoxine hydrochloride (vitamin B6), cyanocobalamin (vitamin B12), DL-alpha-tocopheryl acetate 50% (DL-alpha-tocopheryl acetate, sucrose, caprylic acid) Sodium alkenyl succinate starch, corn starch, water, sodium aluminosilicate), shellac, calcium hydrogen phosphate, edible yellow No. 4, edible yellow No. 5, γ-oryzanol (γ-oryzanol, rice bran powder ), sucrose, silica, inositol, taurine, talc, oxidized starch, gelatin, magnesium stearate, calcium panpolyate, microcrystalline α-cellulose, riboflavin (vitamin B2), palmar wax.
  Arms: EX plus

SUMMARY:
The aim of the present study was to evaluate potential beneficial effects of TTFD® EX PLUS (Prince Pharmaceutical Co., Ltd., Yunlin County, Taiwan) on fatigue and ergogenic functions following physiological challenge. The test used a double-blind crossover design and supplementation for 28 days. 32 male and female 20-30 year-old subjects were divided into two groups in a balanced order according to each individual's initial maximal oxygen uptake and were assigned to receive a placebo with equal gender (non TTFD® EX PLUS with same color/day, n=16, 8 male and 8 female) or TTFD® EX PLUS (600mg/tablet/day, n=16, 8 male and 8 female) every morning. After the intervention, there were 28 days of wash-out, during which time the subjects did not receive further interventions.

ELIGIBILITY:
Inclusion Criteria:

* >20 years old
* >health

Exclusion Criteria:

* No smoking
* drinking habits
* no nutritional supplements or medications
* no food allergies
* normal liver and kidney function
* no diabetes and other chronic diseases

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Exercise endurance exhaustion time | 28 days
  Investigators adopted a double-blind test in which the volunteers, based on their basal maximal oxygen consumption (VO2max). before and after intervention, the individual basal VO2max during pretest was used as a reference to adjust the individually appropriate exercise intensity to measure exhaustive endurance (85% VO2max) and recording the running time from begin to exhaust.
Clinical Biochemistry of lactate level | 28 days
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 5 (E5), 10 (E10), 15 (E15), and 30 (E30) min during the exercise phase, and 20 (R20), 40 (R40), 60 (R60), and 90 (R90) min in the recovery phase. Serum lactate (mmol/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Clinical Biochemistry of ammonia level | 28 days
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 5 (E5), 10 (E10), 15 (E15), and 30 (E30) min during the exercise phase, and 20 (R20), 40 (R40), 60 (R60), and 90 (R90) min in the recovery phase. Serum ammonia (umol/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Clinical Biochemistry of CK level | 28 days
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 5 (E5), 10 (E10), 15 (E15), and 30 (E30) min during the exercise phase, and 20 (R20), 40 (R40), 60 (R60), and 90 (R90) min in the recovery phase. Serum CK (U/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Clinical Biochemistry of glucose level | 28 days
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 5 (E5), 10 (E10), 15 (E15), and 30 (E30) min during the exercise phase, and 20 (R20), 40 (R40), 60 (R60), and 90 (R90) min in the recovery phase. Serum glucose (mg/dL), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Institute of Sports Science, National Taiwan Sport University, Taoyuan District, Taiwan